CLINICAL TRIAL: NCT03583294
Title: A Study on the Uterus, Ovarian and Reproductive Functions According to Conditioning Regimen and Pubertal Status at the Time of Stem Cell Transplantation in a Leukemia Pediatric Population
Acronym: FERTILEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-32; 2017-32 (Other: AP-HM)
Record Dates: First submitted 2018-03-22; First posted 2018-07-11 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-03

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- irradiation regimen before 9 (Experimental): Female who received a hematopoietic stem cell transplantation (HSCT) for AML/CML before 9 years old after conditioning regimen with total body irradation MRI pelvic will be performed
  Interventions: Other: MRI pelvic
- busulfan regimen before 9 (Experimental): Female who received a hematopoietic stem cell transplantation (HSCT) for AML/CML before 9 years old after a busulfan-based conditioning regimen MRI pelvic will be performed
  Interventions: Other: MRI pelvic
- irradiation regimen after 9 (Experimental): Female who received a hematopoietic stem cell transplantation (HSCT) for AML/CML after 9 years old after conditioning regimen with total body irradation MRI pelvic will be performed
  Interventions: Other: MRI pelvic
- busulfan regimen after 9 (Experimental): Female who received a hematopoietic stem cell transplantation (HSCT) for AML/CML after 9 years old after a busulfan-based conditioning regimen MRI pelvic will be performed
  Interventions: Other: MRI pelvic

INTERVENTIONS:
Other: MRI pelvic — Pelvic MRI

SUMMARY:
The French L.E.A. (Leucémie Enfant et Adolescent) program was implemented to prospectively evaluate the long-term health status, quality of life and socio-economic status of childhood acute leukemia (CAL) survivors enrolled in French treatment programs from 1980 to present, in 15 cancer centers. Eligible patients for the study are adult women (≥18 years) from L.E.A. cohort. Project has been approved by the Scientific Advisory Board and the Steering Committee of LEA Cohort. MRI uterus anatomy, follicular ovarian reserve and reproductive function will be assess in 212 adult women who received a hematopoietic stem cell transplantation (HSCT) for CAL. The investigator's objective is to correlate uterus and ovarian function to the conditioning regimen received before HSCT (total body irradiation (TBI) or busulfan - based conditioning) and the pubertal status at the HSCT (before or after puberty).Inclusion period is planned for 2 years. Four patient groups will be compared:

* Group 1: HSCT before nine years and after conditioning regimen with TBI (12 Gy)
* Group 2: HSCT before nine years and after a busulfan-based conditioning regimen
* Group 3: HSCT after nine years and after conditioning regimen with TBI (12 Gy)
* Group 4: HSCT after nine years and after a busulfan-based conditioning regimen

Information will be collected during specific medical visit in one of the investigatory centers. Pelvic MRI and hormonal blood tests will be performed and a medical consultation with a physician specialized in reproductive medicine and oncofertility will be proposed to eligible patients. Data assessed for each women are the following:

* Disease type, age and pubertal status at HSCT, age at evaluation, therapy lines before and after HSCT, conditioning regimen, relapse after HSCT if applicable. Cumulative doses of cyclophosphamide, melphalan, busulfan and radiation will be collected from the LEA database.
* Gynecological characteristics: spontaneous or induced puberty, spontaneous menstrual cycles or Hormone Substitutive treatment (HRT) or amenorrhea without HRT; gestity parity (if pregnancy: spontaneous, after Assisted Reproductive Technologies?), history of ovarian cryopreservation, was information given (and at what age?) about risk of premature ovarian failure and about the gyneco-obstetrical impact of conditioning regimen for HSCT?
* Ovarian follicular reserve: FSH, LH, estradiol, Anti-Müllerian Hormon (AMH) at the day 2-3 of the cycle or whenever if amenorrhea. Ovarian volume and antral Follicle Count will be performed with pelvic sonography.
* Uterine anatomy by MRI, at the end of follicular phase or after estrogen therapy, in order to measure proliferative endometrium. Anatomical parameters will be compare to normal measurements of uterus: uterine volume, myometrial, endometrial and junctionnal zone thickness, cervical length, apparent diffusion coefficient values.
* Reproductive function: spontaneous pregnancy rate or after ART (IVF, oocyte donation), term and mode of delivery, health of the child.

ELIGIBILITY:
Inclusion Criteria:

* Female treated for acute/chronic myeloide leukemia during chidwood and survived from this desease

Exclusion Criteria:

* Female with uneligible MRI exam conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Uterin Anatomy | 1 day
  Pelvic echography: Quantitative estimation of the residual ovarian reserve with the count of antral follicles and the thickness of the endometrium and ovarian volume
  Pelvic IRM: the maximum size of functional endometrium in the proliferative phase

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Courbiere B, Drikes B, Grob A, Hamidou Z, Saultier P, Bertrand Y, Gandemer V, Plantaz D, Plat G, Poiree M, Ducassou S, Pochon C, Dalle JH, Thouvenin S, Paillard C, Kanold J, Sirvent A, Rousset-Jablonski C, Duros S, Gueniffey A, Cohade C, Boukaidi S, Frantz S, Agopiantz M, Poirot C, Genod A, Pirrello O, Gremeau AS, Bringer-Deutsch S, Auquier P, Michel G. The uterine volume is dramatically decreased after hematopoietic stem cell transplantation during childhood regardless of the conditioning regimen. Fertil Steril. 2023 Apr;119(4):663-672. doi: 10.1016/j.fertnstert.2022.12.040. Epub 2023 Jan 7. PMID 36627013